CLINICAL TRIAL: NCT07026279
Title: A Phase 1b/2a, Multicenter, Open Label Study of the Safety, Efficacy and Pharmacokinetics of Narmafotinib in Combination With Modified FOLFIRINOX in Pancreatic Cancer Patients
Brief Title: A Study of Narmafotinib Given in Combination With Modified FOLFIRINOX in Patients With Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amplia Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMP945-PC-202; U1111-1298-5990 (Other: WHO)
Record Dates: First submitted 2025-04-29; First posted 2025-06-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer Metastatic
Keywords: pancreatic cancer; PDAC; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Part A - dose ascending BOIN design Part B - parallel arm (2 dose levels)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Part A is a phase 1b dose-escalation design that will enrol at least 3 participants in each of 4 dose-level cohorts, to determine 2 doses of narmafotinib to be explored in Part B.
  Interventions: Drug: narmafotinib ascending doses
- Part B (Experimental): Part B will determine the efficacy of 2 doses of narmafotinib selected from Part A
  Interventions: Drug: narmafotinib dose comparison

INTERVENTIONS:
Drug: narmafotinib ascending doses — once daily capsules
  Arms: Part A
Drug: narmafotinib dose comparison — once daily capsules
  Arms: Part B

SUMMARY:
This study is testing narmafotinib, a type of drug called a focal adhesion kinase (FAK) inhibitor, when it is given in combination with 4 chemotherapy drugs in a regimen called FOLFIRINOX, to patients who have pancreatic cancer which has metastasised (spread). The study is being run in 2 parts.

Part A will test increasing dose levels of narmafotinib in at least 3 people per dose at up to 4 dose levels to assess safety.

Part B will test 2 of the dose levels from Part A in 20 people per dose, to select the best dose to take forward into future studies.

Participants will take narmafotinib as oral capsules every day. They will also receive mFOLFIRINOX chemotherapy on Day 1 and and Day 15 of 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years at the time of consent.
* Confirmed diagnosis of metastatic pancreatic adenocarcinoma (PDAC) within the 6 weeks prior to study start and have not received treatment for metastatic PDAC.
* Have measurable disease by RECIST v1.1.
* Eligible for treatment with mFOLFIRINOX as standard of care therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
* Have a life expectancy of > 3 months.
* Adequate organ function
* Agree to use effective contraception.

Exclusion Criteria:

* Pregnant or breast-feeding
* Have received any investigational medicinal product (IMP) within 30 days or 5 half-lives (whichever is longer) prior to Day -7.
* Neuroendocrine or acinar cell pancreas tumors.
* Known brain metastases.
* Conditions that could interfere with the swallowing or absorption of study medication.
* Received previous radiotherapy, surgery, chemotherapy, or investigational therapy for the treatment of metastatic disease.
* Received cytotoxic doses of any 5-FU based chemotherapy.
* Any chemotherapy related toxicities greater than grade 1 from prior neoadjuvant or adjuvant therapy for PDAC.
* Human immunodeficiency virus (HIV) infection and/or history of Hepatitis B infection or known to have active hepatitis B or C.
* Uncontrolled angina, myocardial infarction, coronary stenting, stroke, or cerebrovascular accident within 1-year prior to the first dose of study drug.
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis.
* Clinical signs of active infection at the time of Screening or Baseline.
* Clinically significant allergies to narmafotinib, mFOLFIRINOX components (or any of their excipients) that are not likely to be well controlled with pre-medication or other supportive measures.
* Any of the conditions or events outlined in the Contraindications or Special Warnings and Precautions sections of the mFOLFIRINOX component package inserts.
* Peripheral neuropathy > Grade 1.
* Prior treatment with narmafotinib or other FAK inhibitor within the 2 years prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) from Baseline to End of Study | From first dose of study drug to end of study, an expected average of 6 months
  TEAEs during study treatment and follow up periods
Part B: identification of optimal dose of narmafotinib | From first dose of study drug to end of study, an expected average of 6 months
  The optimal dose will be selected based on a review of safety, pharmacokinetics (PK), pharmacodynamics (PD), efficacy, and any other available relevant data

SECONDARY OUTCOMES:
narmafotinib levels in plasma | Days -7, -6, -1, 1 and 15 of Run-In/Cycle 1; and Day 1 of Cycles 2 and 4 (each cycle is 28 days)
  Measurement of maximum concentration (Cmax) of narmafotinib
narmafotinib levels in plasma | Days -7, -6, -1, 1 and 15 of Run-In/Cycle 1; and Day 1 of Cycles 2 and 4 (each cycle is 28 days)
  Measurement of time to Cmax (tmax) of narmafotinib
narmafotinib levels in plasma | Days -7, -6, -1, 1 and 15 of Run-In/Cycle 1; and Day 1 of Cycles 2 and 4 (each cycle is 28 days)
  Measurement of clearance of narmafotinib
Overall response rate (ORR) | Imaging every 56 days per participant, with an expected average duration of 6 months
  ORR based on RECIST 1.1
Overall survival (OS) | Imaging every 56 days per participant, with an expected average duration of 6 months
  OS of participants, defined as time from first dose until death from any cause
Progression free survival (PFS) | Imaging every 56 days per participant, with an expected average duration of 6 months
  PFS of participants, defined as time from first dose to date of first observed progression, based on RECIST, or death from any cause (whichever comes first)
Clinical benefit rate (CBR) | Imaging every 56 days per participant, with an expected average duration of 6 months
  CBR defined as the proportion of patients with complete response (CR) + partial response (PR) + stable disease (SD) with SD for at least 6 months
Duration of response (DOR) | Imaging every 56 days per participant, with an expected average duration of 6 months
  DOR based on RECIST defined as the time from the date of the first confirmed response to the date of progression or death
Disease control rate (DCR) | Imaging every 56 days per participant, with an expected average duration of 6 months
  DCR based on RECIST defined as the proportion of participants who achieve complete response (CR), partial response (PR) or stable disease (SD)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - GenesisCare, St Leonards, New South Wales
  - Epworth Healthcare, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: No